CLINICAL TRIAL: NCT03053310
Title: Determination of the Value of Geriatric Screening to Predict Postoperative Morbidity in an Older Head and Neck Cancer Population (GEROP)
Brief Title: Value of Geriatric Screening to Predict Postoperative Morbidity for Head and Neck Cancer
Acronym: GEROP
Status: Active, not recruiting | Type: Observational
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Johan Abeloos, head of department of maxillofacial surgery, principal investigator, AZ Sint-Jan AV
Other Study IDs: B049201629484
Record Dates: First submitted 2017-02-03; First posted 2017-02-15 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Head and Neck
Keywords: surgery; curative intent; geriatric assessment; 30-day postoperative morbidity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Primary (P) - group: * Patients with a primary diagnosis
  * Patients treated with curative intent (stage I-IVb)
- Relapse (R) - group: * Patients with a recurrent (loco)regional tumour
  * Patients treated with curative intent (stage I-IVb)

SUMMARY:
Background Approximately half of head and neck cancer patients are 65 years or older at diagnosis. Treatment decisions in this older HNCA population are challenging, because of the lack of evidence-based guidelines. Surgery is often the treatment of choice in a HNCA setting where curative treatment is intended. Though chronological age per se has not been reported as a contraindication for surgery, data are limited and often the result of retrospective studies. Measurement of functional age, through a comprehensive geriatric assessment, has been suggested by several international cancer organizations to be a better prognostic indicator. At the divisions of maxillofacial surgery and otorhinolaryngology, a geriatric assessment is part of routine preoperative staging for patients of 70 years old or older.

Objectives The investigators aim to determine the value of G8 to predict 30-day postoperative comorbidity in an older HNCA population undergoing elective curative surgery. Moreover, they aim to examine the vulnerability profile of patients undergoing elective head and neck surgery for an oncology diagnosis.

Study design All patients of 70 years and older, presenting at the divisions of maxillofacial surgery and otorhinolaryngology for curative surgery of a solid head and neck tumour undergo a geriatric consult as part of routine preoperative staging. The presence of postoperative morbidity and mortality within the first 30 days after surgery will be collected as a primary endpoint.

At 30±10 days postoperative, all patients will be re-evaluated with the G8 and the CGA. Patient' quality of life will also be re-examined within 30 days postoperative and again at 6 and 12 months postoperative.

Conclusion There is still no consensus whether older HNCA patients should receive a different treatment compared to younger patients. Data related to the vulnerability profile of older patients requiring HN surgery, and the predictive value of geriatric screening for postoperative morbidity could enable better patient selection in the future.

ELIGIBILITY:
Inclusion Criteria:

* - Patients aged 70 years or older at time of enrolment
* Both female and male patients
* Patients that are Dutch or French-speaking
* Patients with a histologically confirmed malignant tumour in the head and neck region, in specific oral cavity, larynx, and pharynx ('head and neck cancer', defined according to the NCCN guidelines)
* Patients undergoing surgery for a solid head and neck cancer tumour under general anaesthesia. Preoperative data from patients considered ineligible for surgery, will also be registered for scientific purposes
* Patients undergoing surgery and follow-up care at the division of maxillofacial surgery or Department of Otorhinolaryngology, Head and Neck Surgery

Exclusion Criteria:

* - Patients not eligible according to the abovementioned criteria
* Patients with a spinocellular carcinoma of the skin
* Patients with distant metastases (stage IVc)
* Patients with another non-cured cancer, except for a squamous or basal cell carcinoma of the skin
* Patients arriving at the emergency department for urgent surgical intervention
* Patients diagnosed with severe dementia, according to the DSM IV or MMSE ≤18, or diagnosed psychiatric problems impeding proper preoperative assessment

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All consecutive patients, aged 70 years or older, with a primary diagnosis (P-group) or (loco)regional recurrence (R-group) of a solid head and neck tumour, requiring elective surgery under general anaesthesia with curative intent.
Sampling Method: Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2017-01-25 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
30-day postoperative comorbidity | 30 days postoperative

SECONDARY OUTCOMES:
vulnerability percentage of patients undergoing HNCA surgery, based on geriatric consult | at time of surgery
percentage of patients not considered eligible for HNCA surgery, based on geriatric consult and/or MOC consult | prior to surgery, at time of multidisciplinary oncology consult
percentage of patients with major postoperative complications (grade >=3), Graded According to NCI CTCAE Version 4.0 | 30 days postoperative
quality of life, as measured with EORTC questionnaire | 30 days, 6 months and 12 months postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Johan Abeloos, MD, Principal Investigator — AZ Sint-Lucas Brugge
Locations (1):
- AZ Sint-Jan Brugge-Oostende AV, Bruges, Belgium

IPD SHARING:
Plan to Share IPD: No